CLINICAL TRIAL: NCT02414100
Title: Generation of Patient Derived Pancreatic Cancer Cell Lines to Determine Mechanisms of Chemoresistance
Brief Title: Patient Derived Cancer Cell Lines in Identifying Molecular Changes in Patients With Previously Untreated Pancreatic Cancer Receiving Gemcitabine Hydrochloride-Based Chemotherapy
Status: Withdrawn | Type: Observational
Why Stopped: No subjects were enrolled. Study team was not able to grow cell lines for the tumors.
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Other Study IDs: 13C.628; 2013-077 (Other: CCRRC); JT 5543 (Other: JeffTrial Number)
Record Dates: First submitted 2015-03-19; First posted 2015-04-10 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient derived cancer cell lines: Patients receive gemcitabine hydrochloride IV qw 3/4 wk or gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation IV qw 3/4 wk in the absence of disease progression or recurrence per standard of care. Tissue and blood samples are collected for genetic analysis via sequencing.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Cytology Specimen Collection Procedure

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling

SUMMARY:
This pilot research trial studies patient derived cancer cell lines in identifying molecular changes in patients with previously untreated pancreatic cancer and are receiving gemcitabine hydrochloride-based chemotherapy. Cell lines refer to samples taken from the patient's tumor to grow for many months or years in a laboratory, and can therefore be studied scientifically. Studying cell lines in the laboratory may help doctors understand the genetic changes that occur to the tumor during chemotherapy that allows the tumor to resist or grow despite treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the genetic profile of the tumor after progression has occurred, to the tumor prior to treatment.

SECONDARY OBJECTIVES:

I. Additional molecular patterns, beyond genetics, will be analyzed, including ribonucleic acid (RNA) and protein expression.

OUTLINE:

Tissue and blood samples are collected for genetic analysis via sequencing from patients receiving gemcitabine hydrochloride intravenously or gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation. Chemotherapy is not part of the protocol. Per standard of care, patients receive gemcitabine hydrochloride (IV) the first 3 of 4 weeks (qw 3/4 wk) or gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation IV qw 3/4 wk in the absence of disease progression or recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed pancreatic adenocarcinoma, any stage
2. >18 years of age
3. No prior systemic chemotherapy for pancreatic cancer, or currently undergoing first-line treatment for pancreatic cancer, or completed only first-line treatment for pancreatic cancer
4. A plan to undergo gemcitabine-based chemotherapy at Thomas Jefferson or a collaborating institution
5. Abdominal/pelvic CT scan or MRI within 4 months of the study
6. Signed study-specific informed consent

Exclusion Criteria:

1. Pregnancy
2. Prior systemic chemotherapy for pancreatic cancer
3. Gender/Minority/Pediatric Inclusion for Research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treatment naive pancreatic ductal adenocarcinoma (PDA) treated at Thomas Jefferson University or Georgetown University
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Genomic profiles of post-treatment samples with acquired resistance against pre-treatment and germline controls | Up to 5 years
  This method includes a preprocessing step to filter out unreliable reads, a statistical classification step to identify point mutations that differ from both the reference genome hg19 and the control sample at controlled false-positive rate, and a post-processing step to eliminate platform-specific artifacts inherent in next generation sequencing. ANNOVAR software will then be used to analyze candidate point mutations for their predicted impact on protein function, which will be used to select and prioritize specific mutations for validation and/or further study.
Identification of germline mutations in known cancer genes from whole blood genomic deoxyribonucleic acid, and somatic mutations in conditionally reprogrammed cells derived from pre-treatment and post-treatment (e.g., resistant) tumors | Up to 5 years
  The study will be considered a positive study if in any of the patients' samples, unique mutations are identified in the post-treatment derived cell lines that are not present in the pre-treatment derived cell lines from the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Winter, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/